CLINICAL TRIAL: NCT04167891
Title: Comparison of Scores for Early Brain Damage Assessment at Intensive Care Unit Admission After Out of Hospital Cardiac Arrest
Acronym: AfterROSC1
Status: Completed | Type: Observational
Sponsor: AfterROSC (Other)
Responsible Party: Sponsor
Other Study IDs: AfterROSC1
Record Dates: First submitted 2019-11-13; First posted 2019-11-19 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Cardiac Arrest
Keywords: cardiac arrest; hypothermia induced; intensive care unit
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients admitted in the intensive care unit: Patients with return of spontaneous circulation after cardiac arrest regardless of initial rhythm, and admitted in intensive care unit for post cardiac arrest care
  Interventions: Diagnostic Test: Calculation of early prognosis score

INTERVENTIONS:
Diagnostic Test: Calculation of early prognosis score — Early prognosis score will be calculated at intensive care unit admission for each patient based on clinical and biological values as required

SUMMARY:
Even in patients with successful return of spontaneous circulation (ROSC), outcome after cardiac arrest remains poor. The overall in-hospital survival rate widely varies both worldwide and across communities, from 1 to 4 folds according to circumstances of arrest and post-resuscitation interventions. Several studies have already shown that early interventions performed after ROSC, such as treatment of the cause, targeted temperature management, optimal hemodynamic management and extra-corporeal life support in selected patients, could improve the outcome in post-cardiac arrest patients. However, the decision process regarding the allocation of these resources, in parallel with the management of patients' proxies, remains a complex challenge for physicians facing these situations. Consequently, several prediction models and scores have been developed in order to stratify the risk of unfavorable outcome and to discriminate the best candidates for post-resuscitation interventions. Overall, several scores exist, but external validation are lacking and direct comparisons are needed to assess relative interest of scoring systems. Indeed, establishing the optimal scoring system is crucial, for optimal treatment allocation and appropriate information to relatives.

ELIGIBILITY:
Inclusion Criteria:

- All adult patients, major, admitted to intensive care after out-of-hospital cardiac arrest and comatose (defined by Glasgow score ≤ 8) on admission.

Exclusion Criteria:

* cardiac arrest occurring intra-hospital,
* minor patient,
* major patient under guardianship,
* protected persons,
* prior inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is an observational, prospective, multicentric prognostic study. The study period is 1 year, and we plan to include 597 patients in 21 ICUs in France.
  For all patients included, medical history, clinical data, paraclinical results and outcome (at hospital discharge and at 3 months, including modified Rankin score) will be prospectively collected by local investigator, according to an electronical CRF.
Sampling Method: Probability Sample
Enrollment: 1144 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Determination of Area Under Curve of Cerebral Admission Hospital Prognosis (CAHP) Score at intensive care unit admission | Intensive Care Unit Admission (Usually 3 hours after cardiac arrest)
  Determination of AUC for CAHP score as compare to Utstein style criteria.
  CAHP score range from 0 to 300 with higher score indicates poorer prognosis

SECONDARY OUTCOMES:
Determination of Area Under Curve of modified CAHP Score at intensive care unit admission | Intensive Care Unit Admission (Usually 3 hours after cardiac arrest)
  Determination of AUC for modified CAHP score as compare to Utstein style criteria
  mCAHP score range from 0 to 280 with higher score indicates poorer prognosis
Determination of Area Under Curve of simplified CAHP Score at intensive care unit admission | Intensive Care Unit Admission (Usually 3 hours after cardiac arrest)
  Determination of AUC for simplified CAHP score as compare to Utstein style criteria
  sCAHP score range from 0 to 150 with higher score indicates poorer prognosis
Determination of Area Under Curve of OHCA Score at intensive care unit admission | Intensive Care Unit Admission (Usually 3 hours after cardiac arrest)
  Determination of AUC for OHCA score as compare to Utstein style criteria
  OHCA score range from -30 to 60 with higher score indicates poorer prognosis
Determination of Area Under Curve of CREST Score at intensive care unit admission | Intensive Care Unit Admission (Usually 3 hours after cardiac arrest)
  Determination of AUC for CREST score as compare to Utstein style criteria
  CREST score range from 0 to 5 with higher score indicates poorer prognosis
Determination of Area Under Curve of C-Graph Score at intensive care unit admission | Intensive Care Unit Admission
  Determination of AUC for C-Graph score as compare to Utstein style criteria
  C-Graph score range from 0 to 5 with higher score indicates poorer prognosis
Determination of Area Under Curve of TTM Score at intensive care unit admission | Intensive Care Unit Admission (Usually 3 hours after cardiac arrest)
  Determination of AUC for TTM score as compare to Utstein style criteria
  TTM score range from -2 to 35 with higher score indicates poorer prognosis
Determination of Area Under Curve of NULL-PLEASE Score at intensive care unit admission | Intensive Care Unit Admission (Usually 3 hours after cardiac arrest)
  Determination of AUC for NULL-PLEASE score as compare to Utstein style criteria
  NULL-PLEASE score range from 0 to 14 with higher score indicates poorer prognosis
Determination of calibration of each score | Intensive Care Unit Admission (Usually 3 hours after cardiac arrest)
  Determination of calibration of: CAHP, sCAHP, mCAHP, OHCA, CREST, C-Graph, TTM and NULL-PLEASE score

CONTACTS AND LOCATIONS:
Overall Officials: Alain Cariou, MD, PhD, Study Chair — AfterROSC
Locations (27):
- ERASME, Brussels, Belgium
- France (26):
  - CHU Amiens, Amiens
  - CHU Angers, Angers
  - CH Bethune, Béthune
  - CHU Ambroise Paré, Boulogne-Billancourt
  - CH Brive La Gaillard, Brive-la-Gaillarde
  - CH Cherbourg en Cotentin, Cherbourg
  - CHU Créteil, Créteil
  - CHD Vendée, La Roche-sur-Yon
  - CH La Rochelle, La Rochelle
  - CH Versailles, Le Chesnay
  - CH Le Mans, Le Mans
  - CHU Lille, Lille
  - Hospices Civils Lyon, Lyon
  - APHM, Marseille
  - Hopital Privé Jacques Cartier, Massy
  - CHU Montpellier, Montpellier
  - CHRU Nancy, Nancy
  - CHU Nantes, Nantes
  - APHP, CHU Necker, Paris
  - APHP, CHU Saint Louis, Paris
  - Aphp, Hegp, Paris
  - CHU Cochin, Paris
  - CHU Lariboisière, Paris
  - GHP Saint Joseph, Paris
  - Clinique Privé Claude Galien, Quincy-sous-Sénart
  - CH Toulon, Toulon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Renaudier M, Lascarrou JB, Chelly J, Lesieur O, Bourenne J, Jaubert P, Paul M, Muller G, Leprovost P, Klein T, Yansli M, Daubin C, Petit M, Pichon N, Cour M, Sboui G, Geri G, Cariou A, Bougouin W. Fluid balance and outcome in cardiac arrest patients admitted to intensive care unit. Crit Care. 2025 Apr 14;29(1):152. doi: 10.1186/s13054-025-05391-x. PMID 40229890
- [Derived] Lascarrou JB, Bougouin W, Chelly J, Bourenne J, Daubin C, Lesieur O, Asfar P, Colin G, Paul M, Chudeau N, Muller G, Geri G, Jacquier S, Pichon N, Klein T, Sauneuf B, Klouche K, Cour M, Sejourne C, Annoni F, Raphalen JH, Galbois A, Bruel C, Mongardon N, Aissaoui N, Deye N, Maizel J, Dumas F, Legriel S, Cariou A; AfterROSC Network. Prospective comparison of prognostic scores for prediction of outcome after out-of-hospital cardiac arrest: results of the AfterROSC1 multicentric study. Ann Intensive Care. 2023 Oct 11;13(1):100. doi: 10.1186/s13613-023-01195-w. PMID 37819544